CLINICAL TRIAL: NCT01467752
Title: Phase 1 Study for Reconstruction of Metacarpophalangeal Joint Using a Vascularized Cartilage and Bone Graft From the Third Metacarpal
Brief Title: Metacarpophalangeal Joint Reconstruction Using a Vascularized Cartilage and Bone Graft
Acronym: MJRUVCBG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Second Hospital of Qinhuangdao (Other)
Responsible Party: Principal Investigator, Xu Zhang, Director, The Second Hospital of Qinhuangdao
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: XZhang201111; SHQ (Other: the second hospital of qinhuangdao)
Record Dates: First submitted 2011-11-02; First posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Volar Plate Injury, Thumb, Metacarpophalangeal Joint
Keywords: reconstruction; metacarpophalangeal joint; bone graft; MCP joint

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MCP joint (Experimental): reconstruction of metacarpophalangeal (MCP) joint
  Interventions: Procedure: MCP joint

INTERVENTIONS:
Procedure: MCP joint — reconstruction of metacarpophalangeal (MCP) joint using a bone graft
  Other Names: MCP joint reconstruction

SUMMARY:
Traumatic cartilage loss of the joint is central to the development of joint failure in arthritis. The study on the use of a bone graft for reconstruction of metacarpophalangeal joint defects.

DETAILED DESCRIPTION:
The metacarpophalangeal joint is vital for hand function. Cartilage loss of the joint is central to the development of joint failure in arthritis. Although various treatments have been proposed, the management remains a challenging problem.Previous anatomical studies have shown that, at the base of the metacarpal, there were nutrient arteries inserting into the dorsum of the metacarpal. The nutrient arteries arise from the distal and middle dorsal carpal arches that run distally to the first to fourth dorsal metacarpal arteries (DMAs. These studies prompt us to use a reverse vascularized cartilage and bone graft based on the DMA. The metacarpal consists of a widened proximal base. The joint surface to the capitate is convex anteriorly and dorsally concave, where it extends to the styloid process on the dorsolateral aspect of the metacarpal base. The unique contour stimulates our imagination and creativity to use a portion of the joint surface for reconstruction of metacarpophalangeal joint defects. The purpose of this study is to report the novel technique and to evaluate the effectiveness of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. a cartilage defect at either proximal or distal MCP joint;
2. either an acute or old injury;
3. loss of 1/4 of joint entire surface that seen on plain radiographs, CT scan, and intraoperative finding;
4. and with or without MCP joint subluxation.

Exclusion Criteria:

1. large defects involved double joint surfaces;
2. the size of the defect involving less than 1/4 of the joint surface;
3. associate with infection or other diseases that restrict to use the technique.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2005-01; Primary Completion 2005-01 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Range of motion; Arm, Shoulder and Hand questionnaire | 4 years
  The active motions of the hand were measured by a goniometer. The patients rated their MCP joint pain, the donor joint pain, and scar pain using a line by a visual analogue scale (VAS). We used the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire to assess the hand function.

SECONDARY OUTCOMES:
Pain | 4 years
  joint pain is assessed using visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhang, MD, Study Chair — The Second Hospital of Qinhuangdao
Locations (1):
- The second hospital of Qinhuangdao, Qinhuangdao, Hebei, China

REFERENCES:
- [Result] Sebastin SJ, Mendoza RT, Chong AKS, Peng YP, Ono S, Chung KC, Lim AYT. Application of the dorsal metacarpal artery perforator flap for resurfacing soft-tissue defects proximal to the fingertip. Plast Reconstr Surg. 2011 Sep;128(3):166e-178e. doi: 10.1097/PRS.0b013e318221ddfa. PMID 21865990
- See also: Application of the dorsal metacarpal artery perforator flap for resurfacing soft-tissue defects proximal to the fingertip — http://www.ncbi.nlm.nih.gov/pubmed?term=Application%20of%20the%20dorsal%20metacarpal%20artery%20perforator%20flap%20for%20resurfacing%20soft-tissue%20defects%20proximal%20to%20the%20fingertip.